CLINICAL TRIAL: NCT04058366
Title: A Phase 3, Open-label Study Evaluating the Long-term Safety and Efficacy of VX-445 Combination Therapy in Subjects With Cystic Fibrosis Who Are Heterozygous for the F508del Mutation and a Gating or Residual Function Mutation (F/G and F/RF Genotypes)
Brief Title: Study Evaluating the Long-term Safety and Efficacy of VX-445 Combination Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX18-445-110; 2019-000833-37 (EudraCT Number)
Expanded Access: NCT04058210 (Approved for marketing)
Record Dates: First submitted 2019-08-14; First posted 2019-08-15 (Actual); Results first posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2023-12

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — elexacaftor, ivacaftor, tezacaftor drug combination; ivacaftor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ELX/TEZ/IVA (Experimental): Part A: Participants received ELX (elexacaftor) 200 milligram (mg) once daily (qd)/TEZ 100 mg qd/IVA 150 mg every 12 hours (q12h) in the treatment period for 96 weeks.
  Part B: Participants from certain countries participated in Part B and continued to receive ELX 200 mg qd /TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 48 weeks.
  Interventions: Drug: ELX/TEZ/IVA; Drug: IVA

INTERVENTIONS:
Drug: ELX/TEZ/IVA — Fixed-dose combination (FDC) tablet for oral administration.
  Other Names: VX-445/VX-661/VX-770; elexacaftor/tezacaftor/ivacaftor
Drug: IVA — Tablet for oral administration.
  Other Names: VX-770; ivacaftor

SUMMARY:
This study evaluated the long-term safety, efficacy, and pharmacodynamics of elexacaftor (ELX, VX-445) in triple combination (TC) with tezacaftor (TEZ) and ivacaftor (IVA) in subjects with cystic fibrosis (CF) who are heterozygous for the F508del mutation and a gating or residual function mutation (F/G and F/RF genotypes).

ELIGIBILITY:
Key Inclusion Criteria:

* Completed study drug treatment in parent study (VX18-445-104); or had study drug interruption(s) in parent study but completed study visits up to the last scheduled visit of the Treatment Period in the parent study

Key Exclusion Criteria:

* History of study drug intolerance in parent study

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (84):
- United States (33):
  - Banner University of Arizona Medical Center, Tucson, Arizona
  - Miller Children's Hospital / Long Beach Memorial, Long Beach, California
  - Stanford University, Palo Alto, California
  - University of California Davis Medical Center, Sacramento, California
  - University of California San Francisco, Lung Transplant Program, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - University of Miami Miller School of Medicine, Miami, Florida
  - Central Florida Pulmonary Group, PA, Orlando, Florida
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Massachusetts General Hospital Cystic Fibrosis Center Clinical Rsearch Center, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Michigan Medicine, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine / St. Louis Children's Hospital, St Louis, Missouri
  - Mount Sinai Beth Israel, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - UC Health Holmes, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital/University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - ProMedica Toledo Hospital/Toledo Children's Hospital/Pediatric Pulmonary & Cystic Fibrosis Center, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Dell Children's Medical Group, Austin, Texas
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Utah / Primary Children's Medical Center, Salt Lake City, Utah
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Australia (7):
  - The Prince Charles Hospital, Chermside
  - Alfred Hospital, Melbourne
  - Telethon Kids Institute, Nedlands
  - The Royal Children's Hospital, Parkville
  - Mater Adult Hospital, South Brisbane
  - Queensland Children's Hospital, South Brisbane
  - Westmead Hospital, Westmead
- Belgium (4):
  - Cliniques Universitaires de Bruxelles Hopital Erasme, Brussels
  - Universitair Ziekenhuis Brussel - Campus Jette, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
- Canada (2):
  - McGill University Health Center, Montreal
  - St. Paul's Hospital, Vancouver
- Juliane Marie Center, Rigshospitalet, Copenhagen, Denmark
- France (8):
  - Centre Hospitalier Lyon Sud, Benite Cedex
  - Groupe Hospitaler Pellegrin, CHU De Bordeaux, Bordeaux
  - CHRU de Lille - Hopital Albert Calmette, Lille
  - CHU Marseille - Hopital Nord, Marseille
  - CHU de Montpellier - Hopital Arnaud de Villeneuve, Montpellier
  - Hopital Cochin, Paris
  - Hopital Necker, Enfants Malades, Paris
  - Hopital Pontchaillou CHU de Rennes, Rennes
- Germany (6):
  - Charite Paediatric Pulmonology Department, Berlin
  - Ruhrlandklinik Westdeutsches Lungenzentrum am Klinikum Essen, Essen
  - Justus-Liebig-Universitaet Gießen Zentrum fur Kinderheilkunde und Jugendmedizin, Giessen
  - Universitätsklinikum Halle (Saale) / Universitätsklinik und Poliklinik für Innere Medizin, Schwerpunkt Pneumologie, Halle
  - Pneumologisches Studienzentrum Muenchen-West, München
  - University Hospital Wuerzburg, Würzburg
- Ireland (4):
  - Beaumont Hospital, Dublin
  - Children's Health Ireland at Crumlin, Dublin
  - St. Vincent's University Hospital, Dublin
  - University Hospital Limerick (Adults), Limerick
- Italy (5):
  - Azienda Ospedaliero Universitaria Ospedale Riuniti, Ancona
  - IRCCS Istituto Giannina Gaslini-Ospedale Pediatrico, Genova
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale Pediatrico Bambino Gesu, Rome
  - Azienda Ospedaliera di Verona-Ospedale Civile Maggiore, Verona
- Netherlands (2):
  - Academic Medical Center, Amsterdam
  - University Medical Center, Utrecht, Department of Pulmonology and Tuberculosis, Heidelberglaan
- Spain (4):
  - Hospital Universitari Vall d´Hebron Servicio de Broncoscopia, Barcelona
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario y Politecnico La Fe, Valencia
- United Kingdom (8):
  - Papworth Hospital NHS Foundation Trust, Papworth Everard, Cambridge
  - Royal Devon and Exeter NHS Foundation Trust, Royal Devon and Exeter Hospital, Exeter
  - Clinical Research Facility, Queen Elizabeth University Hospital, Glasgow
  - St. James University Hospital, Leeds
  - Liverpool Heart and Chest Hospital, Liverpool
  - Royal Brompton & Harefield NHS Foundation Trust, Royal Brompton Hospital, London
  - Wythenshawe Hospital, Manchester
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent research/clinical-trial-data-sharing.

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted as a single part study (Part A) in countries including United States (US), and the protocol for other countries was amended as a regional protocol so that participants in these countries had the opportunity to participate for up to an additional 48 weeks in Part B.
Pre-assignment Details: Participants from parent study VX18-445-104 (NCT04058353) were enrolled in this study. A total of 251 participants were enrolled in this study.
Period: Overall Study
Arm/Group | ELX/TEZ/IVA
Started | 251
Completed | 215
Not Completed | 36
Not completed — Adverse Event | 14
Not completed — Withdrawal of Consent (not due to AE) | 7
Not completed — Commercial drug is available for participants | 6
Not completed — Death | 1
Not completed — Other non-compliance | 2
Not completed — Other | 6

BASELINE CHARACTERISTICS:
Population: The open label Full Analysis Set (OL-FAS) is defined as all enrolled participants who have received at least 1 dose of study drug in the open-label study.
Groups:
- ELX/TEZ/IVA: Part A: Participants received ELX 200mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 96 weeks.
  Part B: Participants from certain countries participated in Part B and continued to receive ELX 200 mg qd /TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 48 weeks.
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 251
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124
  Male | 127
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 224
  Not collected per local regulations | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 225
  Black or African American | 2
  Other | 5
  Not collected per local regulations | 18
  More than one race | 1

OUTCOME MEASURES:

1. Primary Outcome: Part A: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: From Baseline up to Week 100
Population: The open label (OL) Safety Set for Part A was defined as all participants who received at least 1 dose of study drug in the OLS Part A (participants were assigned based on parent study actual treatment).
Measure: Count of Participants; unit: Participants
Groups:
- Part A: ELX/TEZ/IVA: Participants received ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 96 weeks.
Arm/Group | Part A: ELX/TEZ/IVA
Number analyzed (Participants) | 251
Participants
  Participants with TEAEs | 241
  Participants with SAEs | 38

2. Secondary Outcome: Part A: Absolute Change From Parent Study Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline at Week 96
Population: The OL Full Analysis Set (OL-FAS) for Part A is defined as all enrolled participants who have received at least 1 dose of study drug in the open-label study. This analysis set included study 104 parent study participants who received Control IVA or TEZ/IVA and ELX/TEZ/IVA. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome. Here "Number Analyzed" signifies participants who were evaluable for the specified category.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage points
Groups:
- ELX/TEZ/IVA: All participants who received Control (IVA or TEZ/IVA) or ELX/TEZ/IVA in parent study 104 were to receive ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 96 weeks in Part A of this study.
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 176
percentage points
  Control-IVA or TEZ/IVA: Change at Week 96: number analyzed (Participants) | 80
  Control-IVA or TEZ/IVA: Change at Week 96 | 4.1 [2.5 to 5.7]
  ELX/TEZ/IVA: Change at Week 96: number analyzed (Participants) | 96
  ELX/TEZ/IVA: Change at Week 96 | 3.7 [2.2 to 5.2]

3. Secondary Outcome: Part A: Absolute Change From Parent Study Baseline in Sweat Chloride (SwCl)
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline at Week 96
Population: The OL Full Analysis Set (OL-FAS) for Part A is defined as all enrolled participants who have received at least 1 dose of study drug in the open-label study. This analysis set included study 104 parent study participants who received Control IVA or TEZ/IVA and ELX/TEZ/IVA. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome. Here, "Number Analyzed" signifies participants who were evaluable for the specified category.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimole per liter (mmol/L)
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 186
millimole per liter (mmol/L)
  Control-IVA or TEZ/IVA: Change at Week 96: number analyzed (Participants) | 90
  Control-IVA or TEZ/IVA: Change at Week 96 | -23.0 [-25.8 to -20.1]
  ELX/TEZ/IVA: Change at Week 96: number analyzed (Participants) | 96
  ELX/TEZ/IVA: Change at Week 96 | -22.6 [-25.4 to -19.9]

4. Secondary Outcome: Part A: Absolute Change From Parent Study Baseline in Body Mass Index (BMI)
Description: BMI was defined as weight in kilogram (kg) divided by height in square meter (m^2).
Time Frame: From Baseline at Week 96
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 207
kg/m^2
  Control-IVA or TEZ/IVA: Change at Week 96: number analyzed (Participants) | 97
  Control-IVA or TEZ/IVA: Change at Week 96 | 1.15 [0.84 to 1.45]
  ELX/TEZ/IVA: Change at Week 96: number analyzed (Participants) | 110
  ELX/TEZ/IVA: Change at Week 96 | 0.83 [0.54 to 1.11]

5. Secondary Outcome: Part A: Absolute Change From Parent Study Baseline in BMI Z-score
Description: BMI was defined as weight in kilogram (kg) divided by squared height in meters (m^2). The z-score is a statistical measure to describe whether a value was above or below the standard. A z-score of 0 is equal to the standard. Lower numbers indicate values lower than the standard and higher numbers indicate values higher than the standard.
Time Frame: From Baseline at Week 96
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: z-score
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 18
z-score
  Control-IVA or TEZ/IVA: Change at Week 96: number analyzed (Participants) | 7
  Control-IVA or TEZ/IVA: Change at Week 96 | 0.11 [-0.17 to 0.40]
  ELX/TEZ/IVA: Change at Week 96: number analyzed (Participants) | 11
  ELX/TEZ/IVA: Change at Week 96 | 0.40 [0.17 to 0.62]

6. Secondary Outcome: Part A: Absolute Change From Parent Study Baseline in Body Weight
Time Frame: From Baseline at Week 96
Population: The OL Full Analysis Set (OL-FAS) for Part A is defined as all enrolled subjects who have received at least 1 dose of study drug in the open-label study. This analysis set included study 104 parent study participants who received Control IVA or TEZ/IVA and ELX/TEZ/IVA. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome. Here, "Number Analyzed" signifies participants who were evaluable for the specified category.
Measure: Least Squares Mean (95% Confidence Interval); unit: Kilogram (Kg)
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 207
Kilogram (Kg)
  Control-IVA or TEZ/IVA: Change at Week 96: number analyzed (Participants) | 97
  Control-IVA or TEZ/IVA: Change at Week 96 | 3.6 [2.7 to 4.6]
  ELX/TEZ/IVA: Change at Week 96: number analyzed (Participants) | 110
  ELX/TEZ/IVA: Change at Week 96 | 2.9 [2.0 to 3.8]

7. Secondary Outcome: Part A: Absolute Change From Parent Study Baseline in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: From Baseline at Week 96
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 208
units on a scale
  Control-IVA or TEZ/IVA: Change at Week 96: number analyzed (Participants) | 97
  Control-IVA or TEZ/IVA: Change at Week 96 | 7.2 [4.1 to 10.4]
  ELX/TEZ/IVA: Change at Week 96: number analyzed (Participants) | 111
  ELX/TEZ/IVA: Change at Week 96 | 8.1 [5.1 to 11.1]

ADVERSE EVENTS:
Time Frame: Day 1 through Safety follow-up (up to Week 100 for Part A and up to Week 52 for Part B)
Description: The study was conducted as a single part study (Part A) in countries including United States (US) and the protocol for other countries was amended so that participants in these countries had the opportunity to participate for up to an additional 48 weeks in Part B. The adverse events data has been reported for both the parts separately. MedDRA 24.1 applied for Part A and MedDRA 25.1 applied for Part B.
Groups:
- Part B: ELX/TEZ/IVA: Part B: Participants from certain countries participated in Part B and continued to receive ELX 200 mg qd /TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 48 weeks.
Arm/Group | Part A: ELX/TEZ/IVA | Part B: ELX/TEZ/IVA
All-Cause Mortality (participants affected / at risk) | 1/251 | 0/84
Serious Adverse Events (participants affected / at risk) | 38/251 | 3/84
Other Adverse Events (participants affected / at risk) | 223/251 | 48/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: ELX/TEZ/IVA (N=251) | Part B: ELX/TEZ/IVA (N=84)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Aspergilloma (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Infective exacerbation of bronchiectasis (Infections and infestations) | 2 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 16 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 0
Epididymal cyst (Reproductive system and breast disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: ELX/TEZ/IVA (N=251) | Part B: ELX/TEZ/IVA (N=84)
Abdominal pain (Gastrointestinal disorders) | 13 | 2
Constipation (Gastrointestinal disorders) | 17 | 1
Diarrhoea (Gastrointestinal disorders) | 48 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 13 | 1
Nausea (Gastrointestinal disorders) | 28 | 2
Fatigue (General disorders) | 40 | 0
Pyrexia (General disorders) | 36 | 2
COVID-19 (Infections and infestations) | 52 | 17
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 61 | 17
Nasopharyngitis (Infections and infestations) | 40 | 7
Upper respiratory tract infection (Infections and infestations) | 15 | 6
Vaccination complication (Injury, poisoning and procedural complications) | 28 | 0
Alanine aminotransferase increased (Investigations) | 16 | 0
Aspartate aminotransferase increased (Investigations) | 16 | 0
Blood creatine phosphokinase increased (Investigations) | 26 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 0
Headache (Nervous system disorders) | 71 | 4
Anxiety (Psychiatric disorders) | 28 | 1
Depression (Psychiatric disorders) | 16 | 0
Insomnia (Psychiatric disorders) | 15 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 65 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 20 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 18 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 42 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 17 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 19 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 15 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 34 | 3
Rash (Skin and subcutaneous tissue disorders) | 19 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/66/NCT04058366/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/66/NCT04058366/SAP_001.pdf